CLINICAL TRIAL: NCT06127563
Title: Caring for Frail Patients Through Vaccination
Acronym: CAREVAX
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 5819
Record Dates: First submitted 2023-06-12; First posted 2023-11-13 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-07

CONDITIONS: Vaccination Uptake

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: creation of a clinical pathway to increase vaccination coverage in frail patients — creation of a clinical pathway to increase vaccination coverage for frail patients, integrating hospital and local health units through an automated algorithm

SUMMARY:
The CareVax project aims to find frail patients at Fondazione Policlinico Universitario 'A. Gemelli' IRCCS who could benefit from vaccinations against pneumococcal, Zoster, flu, HBV and SARS-CoV-2. This will reduce hospital stays, long-term effects, and deaths related to these diseases, as outlined in the PNPV (National Plan for Vaccine Prevention) 2017-2019 and Ministry of Health circulars from September, October, December 2022, and January 2023. Eligible patients, upon consent, will be identified by applying an automated algorithm to the patient's electronic health record and vaccination history contained in the regional vaccination registry. Identified patients will be contacted either directly if they are admitted to the inpatient wards of the Fondazione Policlinico Universitario "A.Gemelli" IRCCS (FPG) Hospital, or by messaging or e-mail in the case of access to the FPG for follow-up or routine visits or day hospital or day surgery service. Patients contacted, depending on their frail condition, will be booked for vaccination at an hospital vaccine clinic (extremely vulnerable patients) or a Local Health Unit (ASL Roma1) vaccine clinic respectively (frail patients).

The project envisages a validation phase of the algorithm, through the evaluation of its concordance with the judgement of a blinded clinician on a small group of patients Patients' engagement and a proper communication system with them will be carried through an interoperable digital system aimed at booking the new vaccination appointment, reminding it and providing patients with all the information needed.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or more,
* Patients who have accessed one of the enrolled departments (Dermatology, Oncological gynaecology, Geriatry, Nephrology, Gastroenterology),
* Medical residence in Lazio Region

Exclusion Criteria:

- Patients who do not fulfill 1 or more inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients who have accessed one of the enrolled departments (Dermatology, Oncological gynaecology, Geriatry, Nephrology, Gastroenterology) of teaching hospital A. Gemelli and whose sanitary residence is in Lazio Region (This criteria was inserted because as of now the italian digital infrastructure of the vaccination registry allows easy access only for Regional data) .
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2024-07-17 (Actual); Primary Completion 2026-07-17 (Estimated); Study Completion 2027-07-17 (Estimated)

PRIMARY OUTCOMES:
Vaccinated against influenza at 24 months | 24 months
  Proportion of participants vaccinated against influenza 24 months after the beginning of the study
Vaccinated against influenza at 12 months | 12 months
  Proportion of participants vaccinated against influenza 12 months after the beginning of the study
Vaccinated against influenza at 6 months | 6 months
  Proportion of participants vaccinated against influenza 6 months after the beginning of the study
Vaccinated against COVID19 at 24 months | 24 months
  Proportion of participants fully vaccinated against Covid19 24 months after the beginning of the study
Vaccinated against COVID19 at 12 months | 12 months
  Proportion of participants fully vaccinated against Covid19 12 months after the beginning of the study
Vaccinated against COVID19 at 6 months | 6 months
  Proportion of participants fully vaccinated against Covid19 6 months after the beginning of the study
Algorithm clinician concordance - initial sample of patients | At the start
  Concordance between the clinician's and the algorithm's judgments on patient eligibility for vaccination, measured on a sample of patients.
Algorithm clinician concordance | 24 months
  The proportion of vaccinations confirmed by physicians compared to those proposed by the algorithm.
Feasibility in reaching the patients | 24 months
  Number of patients successfully contacted to offer a vaccination appointment after being considered eligible compared to the number of patients flagged by the algorithm.
Acceptability of the vaccination offer | 24 months
  Number of patients consenting to vaccination appointments compared to the number of patients contacted.
Logistical feasibility of the vaccination pathway | 24 months
  Number of patients presenting to vaccination centers (Hospital or Local Health Authority) compared to the number who have booked a vaccination appointment.
Patients' drop out proportion | 24 months
  Number of patients who drop out or are lost to follow-up versus the total number of patients recruited.

SECONDARY OUTCOMES:
Vaccinated against Hepatitis B virus at 24 months | 24 months
  Proportion of participants vaccinated against Hepatitis B virus 24 months after the beginning of the study
Vaccinated against Herpes Zoster virus at 24 months | 24 months
  Proportion of participants vaccinated against Herpes Zoster virus 24 months after the beginning of the study
Vaccinated against Pneumococcus at 24 months | 24 months
  Proportion of participants vaccinated against Pneumococcus 24 months after the beginning of the study
Vaccinated against Hepatitis B virus at 12 months | 12 months
  Proportion of participants vaccinated against Hepatitis B virus 12 months after the beginning of the study
Vaccinated against Herpes Zoster virus at 12 months | 12 months
  Proportion of participants vaccinated against Herpes Zoster virus 12 months after the beginning of the study
Vaccinated against Pneumococcus at 12 months | 12 months
  Proportion of participants vaccinated against Pneumococcus 12 months after the beginning of the study
Vaccinated against Hepatitis B virus at 6 months | 6 months
  Proportion of participants vaccinated against Hepatitis B virus 6 months after the beginning of the study
Vaccinated against Herpes Zoster virus at 6 months | 6 months
  Proportion of participants vaccinated against Herpes Zoster virus 6 months after the beginning of the study
Vaccinated against Pneumococcus at 6 months | 6 months
  Proportion of participants vaccinated against Pneumococcus 6 months after the beginning of the study
Alerts generated by the algorithm at 24 months | 24 months
  Number of vaccination alerts generated by the algorithm among the study participants in the first 24 months after the beginning of the study

CONTACTS AND LOCATIONS:
Overall Officials: Patrizia Laurenti, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Rome, Lazio, Italy

REFERENCES:
- [Derived] Lontano A, Regazzi L, Tona DM, Di Pumpo M, Porcelli M, Cacciuttolo MG, Parente P, Gasbarrini A, Grandaliano G, Panocchia N, Lopetuso L, Pasciuto T, Cadeddu C, Bruno S, Laurenti P, Pascucci D, Pastorino R. Digital integration between hospitals and local health authorities for enhanced vaccination coverage among frail patients: the CareVax study protocol. Front Public Health. 2025 Jan 30;13:1490244. doi: 10.3389/fpubh.2025.1490244. eCollection 2025. PMID 39949559